CLINICAL TRIAL: NCT00328822
Title: Quetiapine for Primary Insomnia Patients : A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Faculty of Medicine, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: HE490424
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2008-03-18 (Estimated); Status verified 2006-10

CONDITIONS: Primary Insomnia
Keywords: Primary insomnia; Quetiapine; Randomized controlled trial; Double blind
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders | interventions — Quetiapine Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- A (Experimental): Quetiapine
  Interventions: Drug: Quetiapine
- B (Placebo Comparator): Placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Quetiapine
  Arms: A
Drug: placebo
  Arms: B

SUMMARY:
Primary insomnia patients will sleep with Quetiapine not better than without Quetiapine

DETAILED DESCRIPTION:
1. Primary insomnia will be diagnosed according to DSM-IV-TR
2. After consenting, cases will be divided (double blind randomization)in to two arms 2.1 sleep hygiene with placebo group 2.2 sleep hygiene with Quetiapine group
3. outcome measurement: sleep diary, sleep satisfaction visual analog scale and sleep satisfaction likert scale
4. statistical method: dependent T test

ELIGIBILITY:
Inclusion Criteria:

* Primary insomnia Patients by DSM-IV-TR criteria
* cases enrolled: age 18-65 educated

Exclusion Criteria:

* Currently receiving Quetiapine or other hypnotic drugs
* Liver disease
* Patients with heart Dz, Hypertension, thyroid disease
* History of epilepsy or febrile convulsion
* pregnant
* cognitive impairments
* History of Orthostatic Hypotension
* Patient with other Psychiatric conditions or Drug dependence

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2006-12; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
Total Sleep Time | 3 weeks

SECONDARY OUTCOMES:
Sleep Latency Period, Sleep satisfaction | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kanida Tassniyom, MD, Principal Investigator — Department of Psychiatry, Faculty of Medicine, Khon Kaen University
Locations (1):
- Srinagarind Hospital, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

REFERENCES:
- [Derived] Tassniyom K, Paholpak S, Tassniyom S, Kiewyoo J. Quetiapine for primary insomnia: a double blind, randomized controlled trial. J Med Assoc Thai. 2010 Jun;93(6):729-34. PMID 20572379